CLINICAL TRIAL: NCT01345344
Title: Neuroimaging Effects of Cognitive Behavioral Therapy in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Robert Edwards, Robert R. Edwards PhD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2009p001021; R01AR064367 (NIH)
Record Dates: First submitted 2011-04-27; First posted 2011-05-02 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study personnel collecting, entering, and analyzing data are blind to treatment allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive-Behavioral Therapy (Experimental): 8 individual weekly visits with a psychologist for pain-related CBT.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Disease Education (Active Comparator): 8 individual weekly visits with a psychologist for fibromyalgia education (this is an active comparator arm, matched for provider contact).
  Interventions: Behavioral: Disease Education
- Healthy Controls (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Practicing certain cognitive and behavioral pain self-management strategies such as relaxation and changing negative thoughts about pain.
  Arms: Cognitive-Behavioral Therapy
Behavioral: Disease Education — Providing information about fibromyalgia, including its potential causes and management approaches.
  Arms: Disease Education

SUMMARY:
This study design has two components: 1) a cross sectional assessment of brain connectivity and response to pain in healthy controls and demographically matched fibromyalgia patients, and 2) a longitudinal assessment of the same outcomes in fibromyalgia patients randomized to either CBT (Cognitive Behavioral Therapy) or a Disease Education condition.

The investigators will evaluate a group of fibromyalgia patients who will receive CBT treatment once a week for 8 weeks, for a total of 8 treatments. Baseline data from these patients will be compared to results from pain-free controls and a group of education program controls.

Participants will undergo experimental pain assessments as well as brain neuroimaging.

DETAILED DESCRIPTION:
Investigators propose to use fMRI (functional Magnetic Resonance Imaging) to study CNS pain processing during the anticipation and experience of acute pain in individuals with FM and healthy controls. Investigators will recruit patients who are diagnosed with FM as well as healthy controls. After the baseline visit, FM participants will be randomly assigned into the CBT or control condition (Education). Overall, FM Participants will attend 8 treatment visits, and 6 assessment visits (two at baseline, one at mid-treatment, two at the end of treatment, and one at 6 months post-treatment). These assessment visits include a total of 3 fMRI sessions (at baseline, mid-treatment, and end of treatment). Healthy Controls will undergo the same baseline procedures as the FM subjects but will not attend any of the treatment or follow up assessment visits. Findings from this research will provide important information about catastrophizing's CNS (Central Nervous System) correlates.

ELIGIBILITY:
Inclusion Criteria for FM patients:

1. Aged 18-65
2. Female
3. Have a clinical diagnosis of fibromyalgia and meet the Wolfe et al. 2011 research criteria for fibromyalgia
4. On stable doses of medication prior to entering the study and agree not to change medications or dosages (or CAM treatments) during the trial
5. Right-handed
6. Baseline pain intensity of at least 4/10 on average and pain report for at least 50% of days
7. Able to provide written consent

Exclusion Criteria for FM:

1. Comorbid acute pain condition
2. Comorbid chronic pain condition that is rated by the subject as more painful than fibromyalgia
3. Current use of prescription stimulant medications (e.g., modafinil)
4. Routine use of substances of abuse
5. Certain condition that interfere with Quantitative Sensory Testing (QST) and/or fMRI procedures (e.g., Peripheral neuropathy, implanted ferrous metal, claustrophobia etc) or/and any impairment, activity or situation that could prevent satisfactory completion of the study protocol

Inclusion Criteria for Healthy Control Participants

1. Aged 18-65
2. Female
3. Right-handed
4. Able to provide written consent

Exclusion criteria for Healthy Control Participants:

1. Any acute or chronic pain condition (e.g., FM, arthritis)
2. Current use of stimulant medications
3. Routine use of substances of abuse
4. Certain condition that interfere with Quantitative Sensory Testing (QST) and/or fMRI procedures (e.g., Peripheral neuropathy, implanted ferrous metal, claustrophobia etc) or/and any impairment, activity or situation that could prevent satisfactory completion of the study protocol

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical outcome: Brief Pain Inventory (BPI) | Post-treatment, with long-term exploratory outcomes at 6 Months Post-treatment
  Pain-related interference and pain severity
Neurobiological Outcome: Pain Neurocircuitry (fMRI) | Post-treatment
  Bold responses will be assessed with fMRI (3T)

SECONDARY OUTCOMES:
Catastrophizing (PCS) | 4 weeks (mid-treatment), as well as Post-treatment
  Catatrophizing will be assessed with the Pain Catastrophizing Scale (PCS).Investigators hypothesize that early-treatment changes in catastrophizing will produce adaptive brain changes at post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Edwards, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massaschusetts General Hospital, Charlestown, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts

REFERENCES:
- [Derived] Lee J, Protsenko E, Lazaridou A, Franceschelli O, Ellingsen DM, Mawla I, Isenburg K, Berry MP, Galenkamp L, Loggia ML, Wasan AD, Edwards RR, Napadow V. Encoding of Self-Referential Pain Catastrophizing in the Posterior Cingulate Cortex in Fibromyalgia. Arthritis Rheumatol. 2018 Aug;70(8):1308-1318. doi: 10.1002/art.40507. Epub 2018 Jun 22. PMID 29579370